CLINICAL TRIAL: NCT03728816
Title: Multicenter Epidemiologic Study of Severe Community Acquired Pneumonia in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Associate Chief Respiratory Physician, Ruijin Hospital
Other Study IDs: RJ2017NO186-1
Record Dates: First submitted 2018-08-24; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Community-acquired Pneumonia
Keywords: Community Acquired Pneumonia; Epidemiology; Multicenter study
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCAP groups: all the SCAP patients who meet the inclusion criteria

SUMMARY:
This study is aimed to understand the clinical characteristics, etiology and resistance phenotype of major pathogens of SCAP in China through multicenter and prospective investigation. Thus to provide epidemiological basis for improving the SCAP diagnosis and treatment protocol suitable for China.

DETAILED DESCRIPTION:
During the study period, all patients who are diagnosed with SCAP and meet the inclusion criteria in the participating unit should be enrolled in the study . At the end of the trial, each participating unit should complete at least 20 qualified cases, and all participating units should have a total of more than 300 qualified cases.

1. Learn about the etiology of SCAP in China.
2. Grasp the resistance phenotype and molecular epidemiology of major pathogens of SCAP in China.
3. Know the important clinical characteristics of SCAP in China, including age, basic diseases, length of hospital stay, length of stay in ICU, duration of mechanical ventilation, clinical manifestations, imaging findings, complications, mortality, etc.
4. Analyze and clarify the clinical risk factors of affecting SCAP mortality.
5. Understand the current situation of antibiotic treatment of SCAP in China.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yeas;
* Diagnosis of CAP according to the diagnosis and treatment of community-acquired pneumonia in adults: 2016 clinical practice guidelines by the Chinese Thoracic Society, Chinese Medical Association.

Exclusion Criteria:

* Bronchiectasis;
* Active tuberculosis;
* Aspiration pneumonia or obstructive pneumonia;
* Hospitalized in 2 weeks;
* Hospitalized or ventilated ≥5 days;
* Severe immunosuppression patients;
* Irregular follow-up and lost follow-up;
* Withdraw from the study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SCAP patients who meet the inclusion criteria in China
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Microbiological profile of lower respiratory tract specimens | Day 0 of the study
  Record the microbiological profile of lower respiratory tract specimens, including sputum, nasopharyngeal swabs, tracheobronchial aspirates and BAL fluid.
Microbiological profile of urine specimens | Day 0 of the study
  Record the microbiological profile of urine specimens, including all the bacteria explored,especially legionella or streptoccus pneumonia.
Microbiological profile of serum specimens | Day 0,14 days or 21 days of the study
  Record the microbiological profile of serum specimens , including all the bacteria explored, especially legionella, mycoplasma, chlamydia.

SECONDARY OUTCOMES:
General conditions of the participants | Day 0 of the study
  Record the general conditions of the participants when included in the study ,such as demographic , clinical symptoms and signs of the participants, legionella contact history , enrollment date, ICU admitted condition, comorbidities, prior antibiotic treatment and so on.
Inflammatory Parameters | Day 0, 3 days of the study, and until the end of the study(approximately 1 year).
  Record the levels of WBC, CRP, PCT of the participants.
Arterial Blood Gas analysis of the participants | Day 0 of the study
  Record the arterial Blood Gas analysis(pH,PO2,PCO2 etc.) when included in the study.
Chest Image of the participants | Day 0 of the study
  Record the chest radiograph of the participants when included in the study.
Pneumonia Severity Index of the participants | Day 0 of the study
  Record the pneumonia severity index of the participants according to the PSI scoring system,which has been used to decide whether patients with pneumonia can be treated as outpatients or as (hospitalized) inpatients.
CURB-65 Score of the participants | Day 0 of the study
  Assessment of consciousness, urea, respiratory rate, BP, and age 65 years score of the participants(Confusion-1,BUN>7mmol/l-1,Respiratory rate≥30-1，SBP<90mmHg,DBP≤60mmHg-1,Age≥65-1).The risk of death at 30 days increases as the score increases:0-0.6%,1-2.7%,2-6.8%,3-14.0%,4-27.8%,5-27.8%.
Prognosis of the SCAP participants | up to 3 days of the study and until the end of the study(approximately 1 year).
  Record the prognosis(cure,improvement,invalid,recrudesce,death) of the participants through the study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Jieming QU, h.D.,M.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China